CLINICAL TRIAL: NCT02346513
Title: Serum Level of Cobalt and Chromium After Ceramic on Metal Articulation Total Hip Arthroplasty
Acronym: CoM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Won Yong Shon, Professor Won Yong Shon, Department of Orthopedic Surgery, Korea University Guro Hospital, Seoul., Korea University Guro Hospital
Other Study IDs: MD13036
Record Dates: First submitted 2014-11-24; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Hip Replacement Arthroplasty
Keywords: Hip Replacement Arthroplasty; Ceramic on Metal Articulation; Serum level of Cobalt and Chromium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Ceramic on Metal THA: Subgroup A1: Consist of ceramic on metal THAs with short term follow-up (less than 2years)
  Subgroup A2: Consist of ceramic on metal THAs with midterm follow-up (more than 2years)
  Subgroup A3: Consist of bilateral ceramic on metal THAs
  Interventions: Device: Ceramic on Metal Articulation
- B: Non-Ceramic on Metal THA: Patients have THA with non COM bearing
  Interventions: Device: Non-Ceramic on Metal Articulation
- C: Healthy subjects: Patients without any implant or systemic disease, to served as controls

INTERVENTIONS:
Device: Ceramic on Metal Articulation — Patients have THA with ceramic on metal articulation
  Groups: A: Ceramic on Metal THA
Device: Non-Ceramic on Metal Articulation — Patients have THA with non-ceramic on metal articulation
  Groups: B: Non-Ceramic on Metal THA

SUMMARY:
Primary objectives:

1. To measure serum metal ion levels (blood Chromium (Cr) and Cobalt (Co) ion concentration) in patients that received the Ceramic on Metal arthroplasty of hip and who have well functioning primary total hip arthroplasties during short and medium- term follow up time points.
2. To compare blood ion levels of patient that received COM arthroplasty with the blood ion levels of patient receiving non-COM standard total hip arthroplasty (a Metal on polyethylene or ceramic on polyethylene total hip arthroplasty) at short- term and medium-term follow up time points .

Secondary Objective:

1) To determine whether these blood levels correlate with any device specific factors such as: component position, size and type, wear rate and/or patient specific factors such as gender, body mass index, age and activity level.

DETAILED DESCRIPTION:
Peri-prosthetic osteolysis is associated with aseptic loosening of a total hip replacement (THR). It is understood to be a biological response to wear particles, with polyethylene debris thought to be the major cause of the long-term failure.

With total hip replacement (THR) patients now being younger, more active younger, and anticipating much greater longevity, reduced bearing wear becomes increasingly important. Compared to the wear and osteolysis incidence with metal-polyethylene bearings, the historical results of alternate bearings such as metal-on-metal (MOM) and ceramic-on-ceramic (COC) generally showed much lower wear rates and osteolysis was seemingly quite rare. The laboratory wear-rates for metal-metal bearings have generally fallen into the range 1-7 mm3/million cycles (Mc) and 0.1-1 mm3/Mc for run-in and steady-state phases, respectively.

Ceramic-on-ceramic and metal-on-metal bearing surfaces are often employed for total hip replacement because of their resistance to wear. Alternative bearing surfaces such as ceramic-on-ceramic and metal-on-metal eliminate polyethylene wear. Explanted metal-on-metal articulations made of cobalt-chromium-molybdenum (Co-Cr-Mo) alloy have been shown to have extremely low rates of linear wear, and ceramic-on-ceramic bearings even less. A ceramic-on-ceramic articulation was first implanted in 1970 in France. Long-term reports have shown excellent clinical results.

Ceramic-on-ceramic bearings have the advantage of low wear and high biocompatibility. Alumina-ceramic particles are essentially insoluble in organic media and ionisation is therefore unimportant. However, they have some limits: brittleness is a major concern for ceramic, which could lead to clinically relevant failure rates (0.004% head fracture and 0.22% liner fracture. Although Metal-on-metal (MOM) articulations have been seen as one potential solution to the problems associated with UHMWPE-induced osteolysis, metal ions present in the serum and their potential toxic effects both locally and systemically are a cause for concern.

A low wear rate is believed to be critical for extending the implant life of a prosthetic joint, and wear volumes produced by MOM articulations have been estimated to be 40-100 times lower than metal-on-polyethylene bearings. The wear of MOM prostheses is known to be highly dependent upon the materials, tribological design and finishing technique. Clinical studies of retrieved first and second-generation MOM hip prostheses have shown linear penetrations of approximately 5 μm/year. This is equivalent to a wear volume of approximately 1 mm3/year, two orders of magnitude lower than conventional polyethylene acetabular cups.

The observation that a small number of patients with first-generation MOM prostheses exhibited good clinical and radiographical results after 20 years in vivo led to the development of second-generation MOM hip prostheses, and in 1988 the Metasul prosthesis was introduced into clinical practice. This comprised of a cobalt chrome alloy femoral head articulating on a cobalt chrome alloy acetabular cup. Over 200,000 Metasul combinations have been implanted to date. Short-term clinical performance has been encouraging; with low wear rates, and few prostheses requiring revision. However, long-term clinical performance is as yet unknown.

Although MOM hip prostheses produce significantly lower wear rates than conventional UHMWPE-on-metal couples, and lower wear rates than highly crosslinked UHMWPE-on-metal hip prostheses, there are concerns associated with these bearings. Wear particles have been reported to be in the nanometer size range, an order of magnitude smaller than UHMWPE particles. Therefore, despite a lower wear volume than UHMWPE bearings the number of particles produced are estimated to be greater, possibly between one and ten million particles per step. These small particles have the potential to distribute throughout the body via the lymphatic system, with particles found in the lymph nodes, liver, spleen and bone marrow. As MOM hip prostheses are indicated for younger more active patients these particles will be present at these sites for a long period of time, possibly 30-40 years.

Concern has been expressed about the biological response to metal particles released from metal-on-metal couplings. The levels of cobalt and chromium ions have been measured in the blood and serum in patients with successful THR, but information about the possible release of aluminum from ceramic-on-ceramic articulations is lacking.

A better understanding of the influence of the metallurgy and tribology on wear of the component and improved manufacturing technology have allowed the re-introduction of metal-on-metal articulations in total hip replacement. Excellent early clinical outcome has been reported with the new generation of metal-on-metal components. Retrieval studies of previous metal-on-metal bearings and contemporary implants have shown low rate of wear. These hard bearing surfaces are especially promising for young and active patients. Although metal-on-metal bearings produce significantly less wear debris than metal-on-polyethylene bearing surfaces, the debris generated results in the body being exposed to metal ions for prolonged periods. Concerns exist over metal hypersensitivity, osteolysis, chromosomal mutation, carcinogenicity and fetal exposure to high ion levels. These matters require further investigation, particularly the long-term exposure in younger patients and the recognition that some patients may have unusually high ion levels. From tribological studies, joint simulation testing and clinical trials, it has been proposed that the extent of wear can be reduced by using components with a larger diameter with a high carbon content in the alloy (0.2%), well-adjusted clearance for the components, better implant sphericity and lower surface roughness.

Whilst research has shown that high concentrations of nanometre-sized metal wear particles are cytotoxic to human fibroblasts and macrophages in vitro, there are also concerns about the release of metal ions from these small particles, and the potential effect that these ions have on cells and tissues. Elevated ion concentrations have been reported in both the blood and urine of patients with metallic implant components. In addition, contrary to what might be expected, there is no conclusive evidence that ion levels fall in vivo after the bedding in period of the MOM prostheses, during which wear of the prostheses are higher. Cobalt and chromium ions have high toxicity, and there are very real concerns about the effects of sub-lethal doses of metal ions, which have been shown to cause DNA damage. This damage takes the form of chromosome aberrations and chromosome translocations. Over long periods of exposure the worry is that this will lead to the development of certain types of cancer, such as leukaemia and lymphoma. In animal models elevated levels of cobalt, chromium and nickel have been correlated with increased carcinoma rates. However, reports in the literature of malignancies developing after total hip or knee replacement surgery are exceedingly rare. Out of eight epidemiological studies on the relative risk of cancer after TJR, only one study looked specifically at MOM implants. This study did not find an increased risk of cancer development in the subjects receiving MOM hip prostheses compared to those receiving metal-on-polyethylene hip prostheses. However, all the studies to date have been substantially underpowered in terms of patient numbers required to show a difference between the two prosthesis types.

High levels of cobalt and chromium ions are detected in the blood and urine of patients with metal-on-metal (MOM) hip replacement despite, even with these elements are released as a result of wear at the bearing surfaces. The clinical effects of elevated metal ion levels include local tissue reactions, characterized by increases in T and B cells in the tissues surrounding the hip, and are associated with premature failure of the hip. Systemically, one report suggests reduced numbers of CD8-positive T cells. Metal sensitivity is also a potential problem. Metal ions, whether produced secondary to wear debris or via corrosion can initiate a hypersensitivity response. A delayed cell-mediated response, or delayed-type hypersensitivity response can occur, in which cytokines are released by T-lymphocytes and increased activation of macrophages is seen, which may result in T-cell mediated periprosthetic osteolysis. Many metals can initiate a hypersensitivity response, the most common is nickel followed by cobalt and chromium. Therefore, with the well-documented elevation of cobalt and chromium ions in patients with MOM hip implants, there is a theoretical risk of developing hypersensitivity reactions. Recently, an immune response exclusively associated with second-generation MOM hip prostheses, has been described. Histomorphological changes suggest a type of hypersensitivity reaction to the all-metallic implants. The hypersensitivity hypothesis was further strengthened by the observation that these patients experienced early clinical failure at 11-60 months (mean 29 months), and the fact that patients who received a second MOM prosthesis did not experience any relief of symptoms. Conversely, patients who received either metal-on-polyethylene or ceramic-on-polyethylene couples reported that their symptoms completely disappeared. In a control group of patients with joint prostheses not containing cobalt, chromium or nickel these signs of an immunological reactions were absent. Reports of this type of reaction are becoming increasingly common; however, more research is needed in this area. It is not known whether these patients experience prosthesis failure because of a pre-existing metal sensitivity, or whether metal sensitivity develops because of a high wearing bearing and elevated metal ion levels. Theoretically, there would be an increased probability of developing hypersensitivity to elevated metal ion levels, and hence an increased risk of implant failure.

To reduce the effect of these limitations, such as the breakage of the ceramic insert in COM bearing and to reduce ions release in MOM bearing a hybrid coupling of ceramic-on-metal has been proposed. The theoretical advantage of this new coupling might lead orthopedic surgeons to use it indiscriminately.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed an informed consent to this study approved by the Institutional Review Board
2. Is not morbidly obese
3. Is clinically qualified for THA based on physical examination and medical history
4. Has non inflammatory joint disease( osteoarthritis, traumatic arthritis, avascular necrosis ,pelvic fracture, dysplastic variants)
5. Does not have a previous THA or fusion of the hip
6. Pre-operative Harris hip score was below 75 scores
7. Has follow up period that is between 1-2yr or between 2-6yr
8. Surgery was performed by minimal invasive posterior approach by the single surgeon in all groups
9. Standard postoperative care and rehabilitation protocol for both groups (care providers blinded for implant type/ or not)

Exclusion Criteria:

1. Diagnosis of inflammatory joint disease
2. Any current metal hardware
3. Any arthroplasty in any other joint during study follow-up period
4. Pre-operative deranged levels of serum urea, creatinine
5. Severe medical disability limiting ambulation
6. Occupational exposure to cobalt or chromium
7. If they are taking proprietary multivitamins and minerals
8. Chronic steroid or immunosuppressive therapy
9. Metabolic bone disease other than osteoporosis
10. Has plans to relocate to other geographical area before completion of study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population is being drawn for patients seen in the orthopedics department from (April. 2009 -December 2012) patients are selected based on implant type then further selection is based on inclusion and exclusion criteria. Exclusion criteria are specifically selected to exclude any pathologies, or environmental factors that would confound the study population. Once patients are initially selected they are contacted for participation and brought in for screening. Enrollment proceeds until enough patients have been recruited to meet statistical criteria and provide sufficient study power.
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Serum metal ion analysis | 6 months
  Blood sampling will be performed 2 times during follow-up outpatient clinic visits.
  Second sampling is performed 3 months after first sampling.

SECONDARY OUTCOMES:
Wear Measure | 6 months
  A CADD based software POLYWARE (Draftware Inc, CAD viewing and medical image analysis products, Warsaw, Indiana).It is a three-dimensional technique for the measurement of polyethylene wear in metal backed acetabular components. Using a back-lit digitizing tablet, points from AP and Lateral radiographs are captured by AutoCAD software. Custom programming converts the point data into 3D solid models of the prosthesis. The Migration of the Head/cup center points are used to calculate volume displacement.
Radiographic evaluation | 6 months
  Digitalized radiographs of pelvis; standard anteroposterior and lateral oblique radiographs to measure acetabular osteolysis, ante version and abduction angles, a shoot through radiograph to identify impingement and anterior edge loading.
  Standard digitalized radiographs taken at 120% (PiView STAR, version5, Infinitt, Seoul, Korea) will be used for analysis of osteolytic lines in peg zones of femoral component as described by Amstutz and Delee and Charnley zones of the acetabular component.
WOMAC score | 6 months
  Clinical evaluation through a questionnaire and physical examination
Harris Hip score | 6 months
  Clinical evaluation through a questionnaire and physical examination
UCLA activity score | 6 months
  Clinical evaluation through a questionnaire and physical examination
Number of Participants with Adverse Events | 6 months
  1. Infection
  2. Hypersensitivity
  3. Instability
  4. Impingement
  5. Fracture
  6. loosening
  7. Cardiomyopathy
  8. Neurological changes including sensory change( auditory or visual impairment)
  9. Psychological status change( including depression or cognitive impairment,)
  10. Renal function impairment,
  11. Thyroid dysfunction
  12. Noises from the joint(popping, clicking, grinding or squeaking)

CONTACTS AND LOCATIONS:
Overall Officials: Won Yong Shon, Professor, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea